CLINICAL TRIAL: NCT00643734
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Levofloxacin for the Treatment of Mild to Moderate Community-Acquired Pneumonia in Adults
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Trial of Azithromycin SR Compared With Levofloxacin for the Treatment of Mild to Moderate Pneumonia in Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661103
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: azithromycin sustained release; Other: placebo
- 2 (Experimental)
  Interventions: Drug: levofloxacin; Other: placebo

INTERVENTIONS:
Drug: azithromycin sustained release — azithromycin SR 2.0 g by mouth in the form of a slurry for 1 dose
  Arms: 1
Other: placebo — placebo
  Arms: 1
Drug: levofloxacin — 500 mg (two 250 mg capsules) by mouth once daily for 7 days
  Arms: 2
Other: placebo — placebo
  Arms: 2

SUMMARY:
The study was performed to see if a single, 2.0-g oral dose of azithromycin sustained release (SR) was at least as effective as a 7-day regimen of levofloxacin (500 mg once daily) for the treatment of mild to moderate community-acquired pneumonia, and to assess the efficacy and safety of both treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical evidence of mild to moderate community-acquired pneumonia, including cough productive of sputum and a diagnosis of pneumonia, were included.

Exclusion Criteria:

Key exclusion criteria were treatment with any systemic antibiotic of greater than one dose or one combination dose within the previous 7 days, previously diagnosed conditions which tend to mimic or complicate the course and the evaluation of the evaluation process (e.g., bronchiectasis, lung abscess or empyema, active tuberculosis, pulmonary malignancy, cystic fibrosis, post-obstructive pneumonia), hospitalization in the previous 14 days or infection acquired in the hospital, and residents of a long-term care facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2003-04; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
sponsor assessment of clinical response (cure or failure) in the Clinical Per Protocol population | Test of Cure (TOC) visit (Days 14-21)

SECONDARY OUTCOMES:
laboratory abnormalities | Baseline and TOC visit
sponsor assessment of clinical response (cure or failure) in the remaining study populations | EOT visit and TOC visit
sponsor assessment of clinical response by baseline pathogen for the Bacteriological Per Protocol population | EOT visit and TOC visit
investigator assessment of clinical response (cure or failure) in the Clinical Per Protocol population | TOC visit
sponsor assessment of clinical response (cure or failure) in the Clinical Per Protocol population | End of Treatment (EOT) visit (Days 8-11)
bacteriological response on a per pathogen basis for the Bacteriological Per Protocol population | TOC visit
sponsor assessment of clinical response (cure or failure) in the Clinical Per Protocol population | Long-Term Follow-Up (LTFU) visit (Days 28-35)
summary of baseline susceptibilities | Study endpoint
adverse events | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- United States (31):
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, San Luis Obispo, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, Highlands Ranch, Colorado
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Merrit Island, Florida
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Cumberland, Maryland
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Elkhorn, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Rio Rancho, New Mexico
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Yukon, Oklahoma
  - Pfizer Investigational Site, Downingtown, Pennsylvania
  - Pfizer Investigational Site, King of Prussia, Pennsylvania
  - Pfizer Investigational Site, Morrisville, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Dyersburg, Tennessee
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Walla Walla, Washington
  - Pfizer Investigational Site, Menomonee Falls, Wisconsin
- Canada (10):
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
  - Pfizer Investigational Site, Victoriaville, Quebec
  - Pfizer Investigational Site, North Battleford, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Pfizer Investigational Site, Providencia, Santiago Metropolitan, Chile
- India (6):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Vellore, Tamil Nadu
- Lithuania (3):
  - Pfizer Investigational Site, Alytus
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Peru (2):
  - Pfizer Investigational Site, San Isidro, Lima region
  - Pfizer Investigational Site, San Miguel, Lima region
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661103&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Trial%20of%20Azithromycin%20SR%20Compared%20With%20Levofloxacin%20for%20the%20Treatment%20of%20Mild%20to